CLINICAL TRIAL: NCT02534623
Title: Postoperative Quality of Recovery After Transurethral Resection of the Bladder: Spinal Versus General Anesthesia
Brief Title: Postoperative Quality of Recovery After Transurethral Resection of the Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital Zadar (Other)
Responsible Party: Principal Investigator, Nina Sulen, Anesthesiology and Intensive Medicine Specialist, General Hospital Zadar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GHZ trial 001
Record Dates: First submitted 2015-08-15; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Urinary Bladder Neoplasms; Transurethral Resection of the Bladder; Postoperative Recovery
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Anesthesia, Spinal; Anesthesia, General; Bupivacaine; Fentanyl; Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal anesthesia (Active Comparator): Transurethral resection of the bladder performed under spinal anesthesia.
  Interventions: Procedure: Spinal anesthesia; Drug: bupivacaine; Drug: fentanyl
- General anesthesia (Active Comparator): Transurethral resection of the bladder performed under general anesthesia.
  Interventions: Procedure: General anesthesia; Drug: fentanyl; Drug: propofol; Drug: sevoflurane

INTERVENTIONS:
Procedure: Spinal anesthesia
  Arms: Spinal anesthesia
Procedure: General anesthesia
  Arms: General anesthesia
Drug: bupivacaine
  Arms: Spinal anesthesia
Drug: fentanyl
Drug: propofol
  Arms: General anesthesia
Drug: sevoflurane
  Arms: General anesthesia

SUMMARY:
Transurethral resection of the bladder (TURB) is often performed as an outpatient procedure so high-quality postoperative recovery is particularly important. The aim of this study is to compare postoperative quality of recovery after spinal anesthesia (SA) and general anesthesia (GA) for transurethral resection of the bladder.

DETAILED DESCRIPTION:
After written informed consent is obtained seventy patients aged 18-80 years, ASA (American Society of Anesthesiologists) physical status class I-III scheduled for TURB will be randomly assigned to either spinal anesthesia or general anesthesia. Spinal anesthesia will be performed with 12.5 mg of bupivacaine mixed with 25 mcg of fentanyl. General anesthesia will be performed with propofol and fentanyl and maintained with sevoflurane, without use of neuromuscular blocking agents. Quality of Recovery 40 questionnaire (QoR-40) administered before and 24 hours after surgery will be used for assessment of postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Transurethral resection of the bladder
* Age 18 to 80 years
* ASA I-III

Exclusion Criteria:

* Contraindications for spinal anesthesia
* Chronic pain with use of opioids in the last week
* Psychiatric disorders
* Allergy to medications used in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 40 (QoR-40) | 24 hours
  Quality of Recovery 40 questionnaire at 24 hours

SECONDARY OUTCOMES:
Postoperative opioid consumption | 24 hours
  Postoperative opioid consumption over 24 hours
Postoperative pain measured with visual analogue scale | 1,6 and 24 hours
  Postoperative pain measured with visual analogue scale at 1,6 and 24 hours
Patient satisfaction with anesthesia measured with numerical rating scale | 24 hours
  Overall patient satisfaction with anesthesia measured with numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Nina Sulen, MD, Principal Investigator — General Hospital Zadar
Locations (1):
- General Hospital Zadar, Zadar, Croatia

REFERENCES:
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753
- [Background] Catro-Alves LJ, De Azevedo VL, De Freitas Braga TF, Goncalves AC, De Oliveira GS Jr. The effect of neuraxial versus general anesthesia techniques on postoperative quality of recovery and analgesia after abdominal hysterectomy: a prospective, randomized, controlled trial. Anesth Analg. 2011 Dec;113(6):1480-6. doi: 10.1213/ANE.0b013e3182334d8b. Epub 2011 Sep 16. PMID 21926374
- [Background] Barbosa FT, Castro AA. Neuraxial anesthesia versus general anesthesia for urological surgery: systematic review. Sao Paulo Med J. 2013;131(3):179-86. doi: 10.1590/1516-3180.2013.1313535. PMID 23903267
- [Background] Tyritzis SI, Stravodimos KG, Vasileiou I, Fotopoulou G, Koritsiadis G, Migdalis V, Michalakis A, Constantinides CA. Spinal versus General Anaesthesia in Postoperative Pain Management during Transurethral Procedures. ISRN Urol. 2011;2011:895874. doi: 10.5402/2011/895874. Epub 2011 Jul 12. PMID 22084807